CLINICAL TRIAL: NCT03531008
Title: Biomarkers, Health Outcomes and Healthcare Utilization in People With Resistant Focal Epilepsy
Brief Title: Human Epilepsy Project 2: Resistant Focal Seizures Study
Acronym: HEP2
Status: Completed | Type: Observational
Sponsor: Epilepsy Foundation of America (Other)
Collaborators: The Epilepsy Study Consortium (Other); UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: HEP2/TM0020
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Epilepsy; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Biomarkers
Keywords: focal; partial
MeSH Terms: conditions — Epilepsy; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples will be collected at the first visit and the final visit. A third sample may be collected from those participants who experience a seizure-free period of three months or more during the study period. All blood samples will be retained indefinitely, for use in future research. The specific details of future studies are unknown at this time, but will include genomic, proteomic, metabolomic and transcriptome analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment-resistant focal epilepsy: Individuals with treatment-resistant focal epilepsy

SUMMARY:
The HEP2 study is designed to better understand the challenges of living with focal seizures that do not respond to medication, by following 205 people with medication-resistant focal epilepsy over two years to measure changes in health status, healthcare costs, quality of life, and biomarkers of epilepsy severity and treatment response.

DETAILED DESCRIPTION:
The Epilepsy Foundation is launching a partnership, called the Human Epilepsy Project, in collaboration with the Epilepsy Study Consortium. This study (which is called HEP2 for short) is designed to better understand the challenges of living with focal seizures that do not respond to medication. The HEP2 study will follow 200 people with medication-resistant focal epilepsy (with seizures that occur at least 2 times per month) over two years to measure changes in their seizure frequency, treatments used, adverse events experienced, presence of co-morbidities like depression and anxiety, healthcare costs, and quality of life. Blood samples will also be collected in order to look for biomarkers of epilepsy severity and treatment response.

Participants can join the HEP2 study at any one of nine recruiting study centers. These study centers were selected because they are epilepsy centers with track records of conducting high-quality research in epilepsy and efficiently recruiting participants into studies. The designated sites for the HEP2 study are located in New York, California, Minnesota, Connecticut, Pennsylvania, and Tennessee. A participant may enroll in the HEP2 study but continue to receive their standard epilepsy care with their current physician, as long as the participant is willing to share his or her medical records, and travel to the study center for two or three in person visits at the beginning of the study, after the first year, and a final visit after the second year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years and ≤ 65 years at time of enrollment
2. Diagnosed with focal epilepsy with prior vEEG confirmation; if no VEEG confirmation, but in the opinion of the investigator the seizures are definite, the case can be reviewed and adjudicated by the consortium
3. Failure of adequate trials of 4 AEDs, with at least 2 due to failure of seizure control, including current AEDs
4. Have a seizure frequency of ≥ 2 focal seizures/month, including auras, and at least 1 observable seizures/month, that are countable by the subject and/or caregiver for the 3 months prior to enrollment
5. Able to keep a daily seizure diary, either independently or with assistance from a caregiver
6. Able to retrospectively report number of seizures/month for 3 months prior to enrollment
7. Receiving ≥ 1 AED for treatment of seizures

Exclusion Criteria:

1. Patient has a diagnosis of idiopathic ("primary") generalized epilepsy (e.g., juvenile myoclonic epilepsy, absence epilepsy) or mixed focal and generalized (e.g., Lennox-Gastaut syndrome) or non-epileptic seizures within the last 12 months prior to study entry
2. Progressive medical or neurological disorder (brain tumor, AD, PME, etc.)
3. Proven autoimmune etiology
4. Planning pregnancy in the next 12 months
5. Has completed a pre-surgical evaluation and intends to pursue surgery in the near term
6. Resective surgery and/or RNS/VNS in place less than 12 months prior to enrollment
7. Presence of moderate or greater developmental or cognitive delay (e.g., if an adolescent, not in self-contained classroom; if IQ is documented, should be ≥ 70)
8. History of chronic drug or alcohol abuse (misuse or excessive use that interferes with activities of daily living) within the last 2 years
9. Medical, psychiatric or psychosocial condition that would be expected to interfere with the conduct of the study
10. Enrolled in any interventional study that required a blinded portion or involves a non-FDA approved drug or device

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include a cohort of 205 individuals with focal epilepsy who meet the ILAE definition of treatment resistance.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Seizure freedom rates, seizure frequency and degree of disability | 24 Months
  To prospectively quantify seizure frequency over a 24 month period in a cohort of adults with treatment resistant focal epilepsy.

SECONDARY OUTCOMES:
Medication changes | 24 months
  To prospectively quantify medication changes over a 24 month period in a cohort of adults with treatment resistant focal epilepsy.
Healthcare utilization | 24 months
  To prospectively quantify healthcare utilization

OTHER OUTCOMES:
Biomarkers | 24 months
  Although we are not doing these analyses as part of this study, we plan future studies that would include genomics, proteomics, and metabolomics analyses on these samples. We will also make the sample available to other approved researchers upon request and review.

CONTACTS AND LOCATIONS:
Overall Officials: Brandy Fureman, PhD, Principal Investigator — Epilepsy Foundation; Jacqueline French, MD, Principal Investigator — New York University; Ruben Kuzniecky, MD, Principal Investigator — Northwell Health; Daniel Lowenstein, MD, Principal Investigator — University of California, San Francisco
Locations (10):
- United States (10):
  - University of California San Francisco, San Francisco, California
  - Yale Comprehensive Epilepsy Center, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Idaho Comprehensive Epilepsy Center, Boise, Idaho
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - New York University, New York, New York
  - Northwell Health Comprehensive Epilepsy Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Epilepsy Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
No protected health information is stored in the HEP2 database, and participants are tracked using their unique Participant Identifier only. All requests for data and specimen utilization (via collaboration with HEP2 investigators) will be submitted using a standardized form that will be available on the HEP2 website, and will be modeled on those used in the Gene Discovery in Epilepsy project (epi4k.org). These requests will be reviewed by the HEP2 PIs, and agreement to pursue collaborations and sharing of specimens will be based on: 1) strong scientific justification for the proposed collaborative project; 2) attestation by collaborators that all safeguards related to patient confidentiality and distribution of specimens will be upheld; and 3) track record of collaborators.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available for request one year after the database is locked, and will remain available indefinitely.
Access Criteria: All requests for data and specimen utilization (via collaboration with HEP2 investigators) will be submitted using a standardized form that will be available on the HEP2 website, and will be modeled on those used in the Gene Discovery in Epilepsy project (epi4k.org). These requests will be reviewed by the HEP2 PIs, and agreement to pursue collaborations and sharing of specimens will be based on: 1) strong scientific justification for the proposed collaborative project; 2) attestation by collaborators that all safeguards related to patient confidentiality and distribution of specimens will be upheld; and 3) track record of collaborators.
URL: http://www.humanepilepsyproject.org